CLINICAL TRIAL: NCT00913068
Title: Post Operative Analgesia Using the Transverse Abdominal Plan (TAP) Block in Patients Undergoing a Radical Retropubic Prostatectomy (RRP)
Brief Title: Postoperative Pain Control for Prostatectomy
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ricardo Rendon, Dr, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: version 2 July 13, 2009
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lidocaine; Ropivacaine; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP arm (Experimental): in the experimental arm, the procedure will consist of the staff urologist injecting local anesthetic into the anterior abdominal wall bilaterally from the inside of the abdomen at the end of their surgery
  Interventions: Procedure: Transverse Abdominal Plan (TAP)
- standard post operative pain control (Active Comparator): Our current post operative analgesic strategy involves a multi-modal approach, using local injectable anesthetic around the incision and systemic medications (i.e. non-steroidal anti-inflammatories, acetaminophen and break-through doses of opiates). Some of the more common adverse reactions are reparatory depression, sedation, confusion, delirium, nausea, pruritis, constipation, hypotension and bradycardia. Often it is these resulting side effects that extend the length of in hospital rehabilitation, and decrease a patient's overall satisfaction.
  Interventions: Procedure: standard post op pain control

INTERVENTIONS:
Procedure: Transverse Abdominal Plan (TAP) — An injectable anesthetic is introduced to a specific anatomic area where the sensory neurons supplying the operative field.
  Other Names: lidocaine; ropivacaine
  Arms: TAP arm
Procedure: standard post op pain control — opiates
  Other Names: timed assessments for pain and medications
  Arms: standard post operative pain control

SUMMARY:
The researchers propose to investigate a relatively new anesthetic procedure, in order to maximize patient comfort and minimize the use of narcotics after a radical prostatectomy.

DETAILED DESCRIPTION:
Our current post operative analgesic strategy involves a multi-modal approach, using local injectable anesthetic around the incision and systemic medications (i.e. non-steroidal anti-inflammatories, acetaminophen and break-through doses of opiates). As the amount of opiates used can be significant, we have to be aware of their inherent risks. Opiates have an excellent pain control profile, working peripherally by decreasing the amount of neurotransmitters released from neurons involving noxious stimuli, and also in their central processing. Some of the more common adverse reactions are reparatory depression, sedation, confusion, delirium, nausea, pruritis, constipation, hypotension and bradycardia. Often it is these resulting side effects that extend the length of in hospital rehabilitation, and decrease a patient's overall satisfaction.

Thus we propose the use of a relatively new regional anesthetic technique be employed to further decrease the need for opiates in our prostatectomy patients' post-op course, while adequately controlling their pain.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer for radical prostatectomy

Exclusion Criteria:

* chronic pain or opiate use

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Rendon, MD, Principal Investigator — Queen Elizabeth Health Sciences Centre
Locations (1):
- Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: <75, open radical prostatectomy, December 2010 - September 2011. Ketorolac, paralytics, fentanyl, propofol, sevoflurane or isofluroane use was at discretion of anesthetist. Patients requiring spinal or epidural anesthetics, history of chronic pain, chronic opiate use and and need for second general anesthetic within the first 24 h were excluded.
Pre-assignment Details: 16 were excluded before starting the study due to chronic opiate use, or for requiring a secondary general anesthetic
Groups:
- TAP Arm: in the experimental arm, the procedure will consist of the staff urologist injecting percutaneously 20 mg of ropivacaine bilaterally into the anterior abdominal wall . Postoperative pain management same as per standard arm
- Standard Post Operative Pain Control: Injection of saline. Our current post operative analgesic strategy involves a multi-modal approach, using local injectable anesthetic around the incision and systemic medications (i.e. non-steroidal anti-inflammatories, acetaminophen and break-through doses of opiates). Some of the more common adverse reactions are reparatory depression, sedation, confusion, delirium, nausea, pruritis, constipation, hypotension and bradycardia. Often it is these resulting side effects that extend the length of in hospital rehabilitation, and decrease a patient's overall satisfaction.
Period: Overall Study
Arm/Group | TAP Arm | Standard Post Operative Pain Control
Started | 56 | 54
Completed | 48 | 46
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Arm | Standard Post Operative Pain Control | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (6.5) | 60.6 (6.5) | 60.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 56 | 54 | 110
Region of Enrollment [Number; unit: participants]
  Canada | 56 | 54 | 110

OUTCOME MEASURES:

1. Primary Outcome: Total Milligrams of Opiates
Description: mean number of milligrams used postoperatively
Time Frame: 2, 6,12, 24, 48 and 72 hours
Population: In order to achieve a power of 0.9 with a 20% change in pain scores, 40 patients were needed per arm
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | TAP Arm | Standard Post Operative Pain Control
Number analyzed (Participants) | 48 | 46
mg | 5.15 (4.49) | 2.52 (2.91)
Statistical Analysis 1: Comparison: TAP Arm; Test type: Superiority or Other; p = 0.0012, Chi-squared

ADVERSE EVENTS:
Arm/Group | TAP Arm | Standard Post Operative Pain Control
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 0/56 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes